CLINICAL TRIAL: NCT01065948
Title: A Feasibility Study to Assess Critical Aspects of FAS Performance and Safety Over Several Hours
Brief Title: A Feasibility Study to Assess Critical Aspects of Fluorescence Affinity Sensor (FAS) Performance and Safety Over Several Hours
Acronym: FAS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BioTex, Inc. (Industry)
Collaborators: Endocrinoloogy Associates Houston (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FAS-2009-05
Record Dates: First submitted 2010-02-08; First posted 2010-02-10 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: Diabetes
Keywords: subcutaneous glucose monitoring; diabetes; fluorescence; affinity; biosensor; type I Diabetes; type II diabetes
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patients (Experimental)
  Interventions: Device: Subcutaneous glucose monitoring device

INTERVENTIONS:
Device: Subcutaneous glucose monitoring device — monitor interstitial glucose level every 5 min over 4 hours
  Other Names: Fluorescence Affinity Sensor (FAS)

SUMMARY:
The goal of this clinical research study is to learn about a new minimally invasive glucose monitoring device called Fluorescence Affinity Sensor (FAS). In this study, the FAS will be used to determine its effectiveness for glucose monitoring. Researchers want to find out how the device performs at two different body sites (forearm and abdomen) over 4 hours. The safety and comfort level of the device will also be studied.

DETAILED DESCRIPTION:
The FAS glucose monitoring system is a minimally invasive glucose monitoring device which is not yet approved by the FDA. The FAS system will be used in this study to monitor glucose levels during a glucose tolerance test (GTT) performed in Dr.Orzeck practice. The FAS measures glucose levels in skin tissue of the forearm or the abdomen at a depth of less than 1 mm by inserting a small needle-like device. During the 4-hour GTT, the needle-like FAS is left in the skin tissue. The FAS performance has indicated in prior experiments that it is more stable than competitive commercial glucose-sensing devices. Due to its unique design, its glucose response is more accurate, and less affected by certain drugs (such as pain medicine).

ELIGIBILITY:
Inclusion Criteria:

* Female and male patients with Type I and II diabetes requiring injectable insulin from age 18-80.

Exclusion Criteria:

* Patients with fasting glucose concentration larger than 200 mg/dL will be excluded from the study.
* Children under the age of 18 will not be included because Texas state law would not allow such participants to give informed consent on their own.
* Patients who are required to take certain medications including corticosteroids, diuretics, anticonvulsants, birth-control pills, non-steroidal anti-inflammatory drugs (NSAIDs) and certain high-blood pressure medications will be excluded from the study.
* Pregnant women or any patient who cannot participate in an oral glucose tolerance test will also be excluded from the study. Presence of pacemaker or defibrillator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-11; Primary Completion 2012-06 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
examine accuracy of FAS response to glucose changes in subcutaneous tissue (compared to blood glucose concentrations measured with reference method) | 3 months
monitor safety and performance of FAS response in two different body sites (abdomen, forearm) | 3 months

SECONDARY OUTCOMES:
examine insertion site while the FAS is worn, and after seven days of FAS removal | 3 months
assess comfort level during FAS insertion, when worn during normal activities, and during FAS removal | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Dutt-Ballerstadt, Ph.D., Principal Investigator — BioTex, Inc.
Locations (1):
- Practice of Eric Orzeck, MD, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes